CLINICAL TRIAL: NCT06441045
Title: Double Dose of Third-generation EGFR-TKI Plus Intrathecal Pemetrexed Versus Double Dose of Third-generation EGFR-TKI in NSCLC Patients With Leptomeningeal Progression Following the Treatment of Routine Dose of Third-generation EGFR-TKI: a Phase II Randomized, Multicenter Study
Brief Title: Double Dose of Third-generation EGFR-TKI Plus Intrathecal Pemetrexed Versus Double Dose of Third-generation EGFR-TKI in Patients With LM Progression Following the Treatment of Routine Dose of Third-generation EGFR-TKI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SQS2024-175
Record Dates: First submitted 2024-05-03; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Leptomeningeal Metastasis
MeSH Terms: conditions — Meningeal Carcinomatosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Double Dose of Third-generation EGFR-TKI Plus Intrathecal Pemetrexed (Experimental)
  Interventions: Drug: Double Dose of Third-generation EGFR-TKI; Drug: Intrathecal Pemetrexed
- Double Dose of Third-generation EGFR-TKI (Active Comparator)
  Interventions: Drug: Double Dose of Third-generation EGFR-TKI

INTERVENTIONS:
Drug: Double Dose of Third-generation EGFR-TKI — Double Dose of Third-generation EGFR-TKI
Drug: Intrathecal Pemetrexed — Intrathecal Pemetrexed
  Arms: Double Dose of Third-generation EGFR-TKI Plus Intrathecal Pemetrexed

SUMMARY:
We aim to compare the efficacy and safety of double Dose of Third-generation EGFR-TKI Plus Intrathecal Pemetrexed Versus double Dose of Third-generation EGFR-TKI in patients with leptomeningeal progression following the treatment of routine dose of EGFR-TKI,

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years at the time of signing informed consent, both sexes;
* advanced or metastatic NSCLC, TNM stage IV according to the eighth edition of IASLC 2015;
* with EGFR sensitive mutation (exon 19 deletion or L858R mutation), LM progression after conventional doses of three generation EGFR targeted agents (after 1 + 3,2 + 3 or direct 3-generation targeted therapy). There is no limit on the number of chemotherapy lines. The enrolled patients required brain parenchyma and extracranial lesion stable
* ECOG PS score: 0-3
* Normal main organ function, That is, the following criteria are met:

  1. routine blood examination (no blood transfusion within 14 days, no hematopoietic stimulating factor drugs are corrected state): hemoglobin (Hb) 90g / L; Absolute neutrophil count (ANC) 1.5109 / L; Platelet (PLT) 100109 / L; White blood cell count (WBC) 3.0109 / L;
  2. Biochemical examination: alanine transaminotransferase (ALT) and alanine transaminotransferase (AST) 2.5 upper limit of normal (ULN); Serum total bilirubin (TBIL) 1.5 ULN; Serum creatinine (Cr) of 1.5 ULN or creatinine clearance of 50 ml/min; If any liver metastasis, Then, the total bilirubin 3 ULN, ALT and AST 5 ULN; C) Coagulation function: activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time 12 (PT) 1.5 ULN;

  d) Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) 50%;
* If previously treated with chemotherapy, A washout period of at least 21 days between the last chemotherapy dose and enrollment (if the patient does not receive radiotherapy) is required; Patients who treated brain parenchymal metastases with local radiotherapy or surgery before enrollment, Must be completed and fully recovered from the acute toxicity of radiotherapy / surgery. A minimum 14-day washout period is required between the end of radiotherapy and enrollment. A minimum 30-day washout period is required between the end of surgery and enrollment.
* Expected survival of not less than 3 months
* patients can swallow oral medication (if not oral, can be ground by gastric tube)
* Women of childbearing age must have negative pregnancy test (serum or urine) within 14 days before observation period and 3 months after the last administration; for men, they should undergo surgical sterilization or agree to use appropriate contraception during the observation period and 3 months after the last administration of study drug
* patients voluntarily participate and sign an informed consent (or legal agent), expected to have good compliance and able to cooperate with the study according to the protocol requirements.

Exclusion Criteria:

* Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the study program;
* Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS)
* patient with active bacterial infection, fungal infection (intravenous antibiotics required at initiation of study treatment);
* past history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonia requiring steroid therapy, Or any signs of clinically active interstitial lung disease;
* arterial / venous thrombosis events within 6 months prior to enrollment, Such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
* congestive heart failure (NYHA grade> 2); unstable angina pectoris; a myocardial infarction within 3 months prior to signing an ICF; any 12 supraventricular or ventricular arrhythmia requiring treatment or intervention; Mean QTcF> 470ms from 3 ECG recordings
* other systemic malignancies in the last 5 years, (Except for cured skin basal cell carcinoma and cervical situ carcinoma and ovarian carcinoma);
* Use drugs or supplements known to be the main cause of CYP3A4.
* Persons known to be allergic to any test drug or its excipients;
* pregnant, lactating, reproductive patients unwilling to use effective contraception; ●a clear prior history of neurological or psychiatric disorders, including epilepsy and dementia;
* other conditions considered inappropriate by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From date of randomization until the date of death from any cause assessed up to 12 months after the last patient enrollment

SECONDARY OUTCOMES:
Quality of life by using QLC 30 questionnaire | every 4 weeks, from date of randomization until the date of first documented progression or date of death from any cause, whichever came first assessed up to 12 months after the last patient enrollment
  By using QLC 30 questionnaire to investigate the impact of treatment on patients' QoL specifically the physical and neurological function in patients
LM-PFS | From date of randomization until the date of first documented LM progression or date of death from any cause, whichever came first assessed up to 12 months after the last patient enrollment
LM-ORR | From date of randomization until the date of first documented LM progression assessed up to 12 months after the last patient enrollment
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From date of randomization until the date of first documented LM progression or date of death from any cause, whichever came first assessed up to 12 months after the last patient enrollment
  Safety and tolerability
exLM-PFS | From date of randomization until the date of first documented non-LM progression or date of death from any cause, whichever came first assessed up to 12 months after the last patient enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Gen Lin, Principal Investigator — Fujian Provincial Cancer Hospital, Fuzhou, Fujian, China
Locations (1):
- Gen Lin, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No